CLINICAL TRIAL: NCT04360083
Title: Long-term Assessment of Rhône RéPPOP Care for Overweight and Obese Children.
Acronym: LTR
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0285; 2020-A00787-32 (Other: ID-RCB)
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Overweight, Childhood; Pediatric Obesity
Keywords: Pediatric Obesity; Overweight, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overweight and obese children: Overweight and obese children included in RéPPOP care programs between 2007 and 2010.
  Interventions: Other: Collected data from Rhône RéPPOP database; Other: telephonic questionnaire

INTERVENTIONS:
Other: Collected data from Rhône RéPPOP database — BMI Z-scores at the start and the end of RéPPOP care programs.
Other: telephonic questionnaire — Collected data though the telephonic questionnaire : current declared BMI Z-score.

SUMMARY:
Childhood obesity is a major public health issue since it is a risk factor of adulthood obesity, cardiovascular disease, psychological disorders, and other chronic conditions.

RéPPOP is a two year personalized pathway for multidisciplinary care for overweight and obese children, close to patients' homes.

Short and medium-term assessments of Rhône RéPPOP care for overweight and obese children show encouraging results. Long-term assessment is needed to confirm these results.

The present study aims to assess the long-term efficiency of Rhône RéPPOP care for overweight and obese children by comparing BMI Z-scores at the start and the end of RéPPOP care to the current BMI. This data will be collected through a telephonic questionnaire by the scientific manager.

The study's secondary objectives are to evaluate patients and their families' lifestyle changes and to improve RéPPOP practices.

ELIGIBILITY:
Inclusion Criteria:

- All overweight and obese children included in RéPPOP care programs from 01/01/07 to 31/12/10

Exclusion Criteria:

* Refusal to respond to the telephonic questionnaire
* Subjects who withdraw their consent to participate in the study
* Subjects aged under 12 years

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Overweight and obese children included in RéPPOP care programs between 2007 and 2010
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Comparison of BMI Z-scores at the start and the end of RéPPOP care programs to the current BMI Z score. | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Marc NICOLINO, MD, Principal Investigator — Hospices Civils de Lyon, Endocrino-pediatric service, HFME
Locations (1):
- Hospices civils de Lyon, Endocrino-pediatric service, Bron, France